CLINICAL TRIAL: NCT03273790
Title: Effectiveness and Safety of Nivolumab in Advanced/Metastatic Non-Small Cell Lung Cancer (NSCLC) Patients - Retrospective Study of Japanese Real-World Data Through Clinical Chart Review
Brief Title: A Retrospective Study of the Effectiveness and Safety of Nivolumab in Advanced/Metastatic Non-Small Cell Lung Cancer (NSCLC) Patients in Japan
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-9CR
Record Dates: First submitted 2017-09-05; First posted 2017-09-06 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC patients: Initiated Nivolumab treatment at least once from 01 Apr. 2016 through 31 Dec. 2016

SUMMARY:
A Retrospective Study of the Effectiveness and Safety of Nivolumab in Advanced/Metastatic Non-Small Cell Lung Cancer (NSCLC) Patients in Japan

ELIGIBILITY:
Inclusion Criteria:

* Previously treated advanced/metastatic NSCLC patients treated with nivolumab at least once from 01-Apr-2016 through 31-Dec-2016

Exclusion Criteria:

Patients who meets the inclusion criteria will be included in the analysis to describe real-world clinical usage of nivolumab. However, patients treated with nivolumab falling in following criteria will be excluded for analysis for the other primary endpoint; overall effectiveness:

* History of participation in any clinical trials prior- or post-nivolumab treatment
* Patients who are a part of a Post-marketing surveillance study

Other protocol defined inclusion/exclusion criteria could apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously treated advanced/metastatic NSCLC patients treated with nivolumab in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 939 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Description of clinical usage of nivolumab in previously treated NSCLC patients | Approximately 9 months
Overall Survival (OS) | Approximately 9 months
  Measured from time of initial diagnosis and treatment with nivolumab until date of death
Progression Free Survival (PFS) | Approximately 9 months
  Time since index date (initial diagnosis and treatment with nivolumab) to either the first disease progression date or last known tumor assessment date, or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Percentage of patients receiving bi-weekly nivolumab | Approximately 9 months
Percentage of patients receiving monotherapy or combination therapy | Approximately 9 months
Percentage of patients receiving nivolumab as second or later line of therapy | Approximately 9 months
Median treatment duration and range by line and histology | Approximately 9 months
Rate of permanent and temporary discontinuations | Approximately 9 months
Reasons for discontinuation of nivolumab | Approximately 9 months
Reasons for re-challenge of nivolumab | Approximately 9 months
Objective Response Rate (ORR) as assessed by investigator | Approximately 9 months
  ORR is defined as the number of participants with best overall response (OR) of confirmed complete response (CR) or partial response (PR) divided by the total number of participants who received treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Minato-ku, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm